CLINICAL TRIAL: NCT05740254
Title: Early vs. Late Time-Restricted Eating in Adolescents With Obesity (EL TREA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Alaina P. Vidmar, MD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-22-00395
Record Dates: First submitted 2023-02-08; First posted 2023-02-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Obesity; Time Restricted Feeding; Time Restricted Eating
Keywords: Obesity; Intermitted-fasting; Time Limited Eating
MeSH Terms: conditions — Pediatric Obesity; Intermittent Fasting; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time Restricted Eating (Experimental): early-day TRE (7:00 to 15:00 h)
  Interventions: Behavioral: Early Time Restricted Eating
- Late Time Restricted Eating (Experimental): late TRE (12:00 to 20:00 h)
  Interventions: Behavioral: Late Time Restricted Eating

INTERVENTIONS:
Behavioral: Early Time Restricted Eating — Early Time Restricted Eating 7 AM to 3 PM
  Arms: Early Time Restricted Eating
Behavioral: Late Time Restricted Eating — Late Time Restricted Eating 12 PM to 8 PM
  Arms: Late Time Restricted Eating

SUMMARY:
Determine the effectiveness of how limiting the time you eat within an early or late eating window and fasting for remainder of the day will impact weight loss and body mass index (BMI).

DETAILED DESCRIPTION:
In adults, there is growing evidence that early TRE is more effective in improving metabolic outcomes than other forms of TRE, however it is unclear whether adolescents will be able to adhere to such recommendations. Hence, in the present study we propose a 24-week, 2-arm, parallel randomized pilot trial in 100 adolescents (age 13-18 years, all gender expressions, anticipate 65% Latino) with obesity, to test the preliminary efficacy of early vs. late TRE on glycemic profiles, weight loss, and body composition. We hypothesize that, among adolescents who can adhere to the meal timing recommendations, early TRE will result in greater improvement in metabolic endpoints than late TRE. We will test the hypothesis with 3 specific aims: Aim 1: Test the effect of early vs. late TRE on glycemic profiles and β-cell function. Aim 2: Test the effect of early vs. late TRE on obesity and body composition, and cardiometabolic risk factors. Aim 3: Test the effect of early vs. late TRE on exploratory outcomes including sleep, physical activity, and dietary intake to explore how meal timing may influence occurrence, timing, and distribution of sleep and movement as well as dietary intake and caloric distribution. This study is the first study evaluating the effectiveness of early vs. late TRE in adolescents with obesity at risk for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years with obesity (BMI>95th percentile)
* participant must be willing and able to adhere to the assessments, visit schedules, and eating/fasting periods
* baseline eating window greater than 12 hours.

Exclusion Criteria:

* diagnosis of Prader-Willi Syndrome, brain tumor, or diabetes serious intellectual disability
* previous diagnosis or subthreshold symptoms of an eating disorder (anorexia nervosa, bulimia nervosa, binge-eating disorder)
* parent/guardian-reported physical, mental of other inability to participate in the assessments
* previous bariatric surgery
* current participation in other interventional weight loss studies.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in weight in excess of the 95th percentile at week 24 compared to baseline | week 24
  Change in weight in excess of the 95th percentile

SECONDARY OUTCOMES:
Mean change in total body fat mass as measured on DEXA scan at week 24 compared to baseline | week 24
  Change in total body fat mass measured on DEXA scan
Mean change in percent time in range as captured on contiguous glucose monitor at week 24 compared to baseline | week 24
  %TIR captured on CGM
Mean change in hemoglobin A1c at week 24 compared to baseline | week 24
  HgA1c measured at baseline and week 24
Mean change in ALT at week 24 compared to baseline | week 24
  ALT measured at baseline and week 24
Mean change in systolic and diastolic blood pressure at week 24 compared to baseline | week 24
  Measured systolic and diastolic blood pressure at baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Vidmar, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Clinical characteristics data will be available in CSV format, and will not require the use of specialized tools to be accessed. To facilitate interpretation of the data, study protocol and clinical data dictionary will be shared and associated with the relevant datasets. Information about our research process, including the details of biochemical assays be maintained contemporaneously. This information will be accessible to all members of the research team and will be shared alongside our data. Data to be shared will be made available at the time of associated publication or by the close of the reward. Data will be made available, at minimum, for length of the grant + 5 years. Restrictions on subsequent access, distribution, or reuse of scientific data from this project include confidentiality protections. All data shard will be de-identified and not include any sensitive information or potentially identifying variables.